CLINICAL TRIAL: NCT04974801
Title: A Randomized Cross Over Clinical Trial Assessing the New Provox Life System for Pulmonary Rehabilitation and Quality of Life After Total Laryngectomy
Brief Title: Assessment of the New Provox Life System for Pulmonary Health and Quality of Life After Total Laryngectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atos Medical AB (Industry)
Collaborators: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Prot_Id_3523
Record Dates: First submitted 2021-07-06; First posted 2021-07-23 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Laryngectomy
Keywords: Pulmonary rehabilitation; Quality of Life; Heat and Moisture Exchangers

STUDY DESIGN:
Intervention Model Description: Single center, randomized, prospective crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provox Life HMEs followed by Usual Care HMEs (Other): Use of Provox Life devices during a period of six weeks followed by use of Usual Care devices during a period of six weeks.
  Interventions: Device: Provox Life; Device: Usual Care
- Usual Care HMEs followed by Provox Life HMEs (Other): Use of Usual Care devices during a period of six weeks followed by use of Provox Life devices during a period of six weeks.
  Interventions: Device: Provox Life; Device: Usual Care

INTERVENTIONS:
Device: Provox Life — Use of Provox Life range of HMEs for different situations and their attachments (adhesives and laryngectomy tubes)
Device: Usual Care — Continued Usual Care routines.

SUMMARY:
Background: The benefits of using Heat and Moisture Exchangers (HMEs) for pulmonary rehabilitation after total laryngectomy are widely known. However, current available HMEs do not reach the level of humidification capacity of the nose, and patients adherence to using an HME 24/7 is not always possible. Provox Life HMEs and attachments are a new range of HMEs and attachments, with improved humidification/breathability performance, and designed to suit different situations.

Purpose and aim: In this clinical trial, the new Provox Life System was assessed for pulmonary rehabilitation and QoL after total laryngectomy, and compared with currently available HMEs and attachments.

Methods: Forty laryngectomized patients, who were previous users of HMEs, were randomized to Usual Care or Provox Life for 6 weeks, after which a cross-over occurred. Data was collected at baseline, and after the end of each study period. Additionally, patients filled in a diary and tally sheet to record their forced expectorations and coughing.

ELIGIBILITY:
Inclusion Criteria:

* Total laryngectomy, irrespective of pharynx reconstruction method
* 18 years or older
* Provox XtraHME user
* Provox Adhesive user
* Longer than 3 months after total laryngectomy
* Longer than 6 weeks after postoperative radiotherapy

Exclusion Criteria:

* Medical problems prohibiting the use of HME or adhesive
* Active recurrent or metastatic disease (medical deterioration)
* Recent pulmonary infections/unstable pulmonary condition
* Reduced mobility of arms and/or hands, unable to remove an HME
* Unable to understand the Patient Information and/or unable to give Informed Consent
* Insufficient cognitive ability to handle the HME or adhesive
* LaryButton users

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Average number of forced mucus expectorations per 24 hours | during week 6 of period 1 and period 2 (each period is 6 weeks)
  Patient reported, recorded by Tally sheeting on 3 days

SECONDARY OUTCOMES:
Average number of (involuntary) dry coughs per 24 hours | during week 6 of period 1 and period 2 (each period is 6 weeks)
  Patient reported, recorded by Tally sheeting on 3 days
Coughing Symptoms (COUS) domain score of CASA-Q | Baseline, at the end of period 1, at the end of period 2 (each period is 6 weeks)
  Cough Symptoms (COUS), assessed with validated Coughing and Sputum Assessment Questionnaire (CASA-Q) questionnaire. CASA-Q score between 0-100, with higher scores meaning less symptoms and less impact.
Coughing Impact (COUI) domain score of CASA-Q | Baseline, at the end of period 1, at the end of period 2 (each period is 6 weeks)
  Cough Impact (COUI), assessed with validated Coughing and Sputum Assessment Questionnaire (CASA-Q) questionnaire. CASA-Q score between 0-100, with higher scores meaning less symptoms and less impact.
Sputum Symptoms (SPUS) domain score of CASA-Q | Baseline, at the end of period 1, at the end of period 2 (each period is 6 weeks)
  Sputum Symptoms (SPUS), assessed with validated Coughing and Sputum Assessment Questionnaire (CASA-Q) questionnaire. CASA-Q score between 0-100, with higher scores meaning less symptoms and less impact.
Sputum Impact (SPUI) domain score of CASA-Q | Baseline, at the end of Period 1, at the end of Period 2 (each period is 6 weeks)
  Sputum Impact (SPUI), assessed with validated Coughing and Sputum Assessment Questionnaire (CASA-Q) questionnaire. CASA-Q score between 0-100, with higher scores meaning less symptoms and less impact.
Peristomal skin irritation | Baseline, at the end of Period 1, at the end of Period 2 (each period is 6 weeks)
  Recorded by study specific questionnaire on frequency of Skin irritation.
Average number of days with skin irritation | during week 5 and week 6 of period 1 and period 2 (each period is 6 weeks)
  Patient reported, recorded by daily diary keeping the last two weeks of each study period
Quality of Life by EQ-5D-5L | Baseline, at the end of Period 1, at the end of Period 2 (each period is 6 weeks)
  Patient reported, the descriptive system assesses health in five dimensions, from which a health state index score is calculated, range from 0 to 1, with higher scores indicating higher health utility
Frequency of using sleeping medication | Baseline, at the end of Period 1, at the end of Period 2 (each period is 6 weeks)
  Study-specific questionnaire on use of sleeping medications
Average number of hours of HME use per 24 hours | during week 5 and week 6 of period 1 and period 2 (each period is 6 weeks)
  Patient reported, recorded by daily diary keeping the last two weeks of each study period
Situational usage pattern of Provox Life HMEs | Baseline, at the end of Period 1, at the end of Period 2 (each period is 6 weeks)
  Study-specific questionnaire about the situational use of devices
Patient satisfaction with the Provox Life devices | At the end of Period 1 (Group A), at the end of Period 2 (Group B) (each period is 6 weeks)
  Patient satisfaction with devices through study specific questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Parilla, Dr., Principal Investigator — Universita Cattolica del Sacro Cuore di Roma, Faculty of Medicine and Surgery 'Agostino Gemelli'
Locations (1):
- Universita Cattolica del Sacro Cuore di Roma, Faculty of Medicine and Surgery 'Agostino Gemelli', Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Longobardi Y, Galli J, Di Cesare T, D'Alatri L, Settimi S, Mele D, Bussu F, Parrilla C. Optimizing Pulmonary Outcomes After Total Laryngectomy: Crossover Study on New Heat and Moisture Exchangers. Otolaryngol Head Neck Surg. 2022 Dec;167(6):929-940. doi: 10.1177/01945998221086200. Epub 2022 Mar 22. PMID 35316144